CLINICAL TRIAL: NCT03975140
Title: The Preventive Value of Acupoint Sensitization Based on Stable Angina Pectoris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Sun Xin, the Director of Chinese Evidence-based Medicine Center, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 81590955
Record Dates: First submitted 2019-05-24; First posted 2019-06-05 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: The Clinical Value of Acupoint Sensitization

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypersensitive acupoint group (Experimental)
  Interventions: Procedure: Hypersensitive acupoint group
- Hyposensitive acupoint group (Active Comparator)
  Interventions: Procedure: Hyposensitive acupoint group

INTERVENTIONS:
Procedure: Hypersensitive acupoint group — The first five acupoints in the sensitization sequence were pressed using the traditional Chinese medicine acupoint pressing technique, and each acupoint was pressed for two minutes.
  Arms: Hypersensitive acupoint group
Procedure: Hyposensitive acupoint group — The last five acupoints in the sensitization sequence were pressed using the traditional Chinese medicine acupoint pressing technique, and each acupoint was pressed for two minutes.
  Arms: Hyposensitive acupoint group

SUMMARY:
This study, taking stable angina pectoris as a research carrier, aims to explore the preventive value of acupoint sensitization by conducting a double-blind multi-center randomized controlled trial to compare the effect of stimulating acupoints with different sensitivity on the prevention of angina pectoris.

After the inclusion of eligible patients, the pressure-pain threshold of disease-related acupoints will be detected by using Von Frey detector. Then, the patients will be randomly divided into experimental group and control group. The patients in experimental group will be given acupoints pressure on the five acupoints with the lowest pressure-pain threshold, while the patients in control group will be given acupoints pressure on the five acupoints with the five acupoints with the highest pressure-pain threshold. The two groups will be treated with acupoints pressure 12 times within 4 weeks. The patients will be evaluated three times at baseline, the end of treatment and four weeks after the end of treatment respectively, including angina attack frequency, CCS classification and SAQ score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina pectoris and symptoms of chest pain
* The duration of onset was more than 3 months, and the number of angina attacks in the past month was not less than 2
* Not younger than 35 years old and not older than 80 years old
* Patients will participate in the study voluntarily and have signed the informed consent

Exclusion Criteria:

* Patients with mental retardation
* Patients were contraindicated or unable to complete acupoint sensitization test
* Patients with cardiovascular, digestive, urinary, respiratory, blood, nervous, endocrine system and other serious primary diseases
* Patients with bleeding, allergy constitution
* Patients with abnormal skin or peripheral nerve sensation, abnormal pain sensation, skin ulceration at the sensitization detection site
* Patients with unsatisfactory clinical treatment of hypertension and diabetes

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Change of the number of angina attacks | Change from baseline to week 8
  Change of the number of uncomfortable events that met the criteria for angina in study period

SECONDARY OUTCOMES:
Change of the Canadian Cardiology Society (CCS) Classification of Angina Pectoris | Change from baseline to week 8
  According to the patient's own condition scale, the patients were divided into 4 grades, the mildest being grade I and the most serious being grade IV
Change of the Seattle Angina Questionnaire(SAQ) Score | Change from baseline to week 8
  The maximum score of the scale was 100, and the higher the score, the better the quality of life and the functional state of the patients
Change of the use of Therapeutic Nitroglycerin Drugs | Change from baseline to week 8
  Change of the number of times that patients temporarily took nitroglycerin for angina attacks

CONTACTS AND LOCATIONS:
Locations (1):
- The West China Hospital of Sichuan university, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Huang S, Li L, Liu J, Li X, Shi Q, Li Y, Liu Y, Li M, Ma L, Ning L, Liao X, Ying X, Cai W, Yang F, Wang T, Guo R, Ma W, Chen W, Chen J, Sun X. The Preventive Value of Acupoint Sensitization for Patients with Stable Angina Pectoris: A Randomized, Double-Blind, Positive-Controlled, Multicentre Trial. Evid Based Complement Alternat Med. 2021 Nov 2;2021:7228033. doi: 10.1155/2021/7228033. eCollection 2021. PMID 34765004